CLINICAL TRIAL: NCT03332849
Title: A Phase 1, Multiple Ascending Dose Glucose Clamp Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of HM12470 in Comparison to Insulin Glargine in Subjects With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Multiple Ascending Dose Study of HM12470 in Type 1 and Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM-INS115-103
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Type1 Diabetes Mellitus; Type2 Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): T1DM: Multiple dose subcutaneous administration
  Interventions: Biological: HM12470
- Cohort 2 (Experimental): T1DM: Multiple dose subcutaneous administration
  Interventions: Biological: HM12470
- Cohort 3 (Experimental): T2DM: Multiple dose subcutaneous administration
  Interventions: Biological: HM12470
- Cohort 4 (Experimental): T2DM: Multiple dose subcutaneous administration
  Interventions: Biological: HM12470

INTERVENTIONS:
Biological: HM12470 — HM12470 is a long-acting insulin analogue

SUMMARY:
This is a phase 1 multiple ascending dose (MAD) study, conducted in subjects with Type 1 and Type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* T1DM or T2DM
* Female subjects must be non-pregnant and non-lactating

Exclusion Criteria:

* Pregnant or lactating women
* Participation in an investigational study within 30 days prior to dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 month
  An adverse event is any undesirable and unintended medical event occurring to a subject in a clinical study, whether or not related to the investigational products.

SECONDARY OUTCOMES:
Cmax of HM12470 | 1 month
  - Maximum concentration of HM12470 over the entire dosing period
AUC of HM12470 | 1 month
  - Area Under the Curve of HM12470 over the entire dosing period

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Investigative Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided